CLINICAL TRIAL: NCT01235403
Title: A Multicenter, Open Label Study to Evaluate the Tolerability, Safety and Efficacy of Lacosamide (200mg - 400mg/Day) as add-on Therapy for Patients With Partial Onset Epilepsy Using a Flexible Dose-escalation Schedule and Individualized Maintenance Doses
Brief Title: Trial to Assess Optimized Dosage of Lacosamide as add-on Therapy in Patients With Partial Onset Seizure
Acronym: SELF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP1007; 2010-019268-35 (EudraCT Number)
Record Dates: First submitted 2010-11-03; First posted 2010-11-05 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-03

CONDITIONS: Partial Epilepsies
Keywords: Epilepsy treatment.; Anti-epileptic drugs; Seizures
MeSH Terms: conditions — Epilepsies, Partial; Seizures | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Flexible dosing between 200mg/day and 400mg/day
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide : 50 mg tablets bid. Titration phase: (12 weeks) 100 mg/day: duration 1 to 3 weeks. Then uptitration to optimal therapeutic dose of 200 mg/day to 400 mg/day, in steps of 100 mg/day and a time period per step of 1 to 3 weeks.
  Maintenance phase (12 weeks): Optimal therapeutic dose 200 mg/day to 400 mg/day.
  Taper phase if needed: 3 to 4 weeks
  Other Names: Vimpat®

SUMMARY:
To evaluate if a flexible dose escalation of lacosamide, up to the maximum approved dose of 400 mg/day, or to a clinically effective lower dose for an individual patient, improves the tolerability and safety of lacosamide (200 mg to 400 mg/d) as add-on treatment for patients with partial onset epilepsy.

Explanation of acronym: SELF = Safety Efficacy Lacosamide Flexibility

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of partial-onset epilepsy with or without secondary generalization
* Currently taking 1 to 3 concomitant marketed antiepileptic drugs
* 18 years and older at study entry

Exclusion Criteria:

* Previous use of lacosamide
* Hypersensitivity to any component of lacosamide
* Patients with partial onset seizures not clearly identifiable
* History of generalized epilepsy
* History of status epilepticus within last 12 months
* Uncountable seizures due to clustering within last 12 weeks
* Non epileptic events, including pseudoseizures, conversion disorder that could be confused with seizures
* History of drug or alcohol abuse
* History of suicide attempt
* Progressive cerebral disease
* Concomitant treatment of felbamate
* Prior or concomitant vigabatrin use
* Under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (32):
- France (32):
  - Amiens
  - Aubenas
  - Auxerre
  - Bordeaux
  - Brest
  - Caen
  - Carpentras
  - Châteaubriand
  - Colmar
  - Créteil
  - Gap
  - Gonesse
  - La Rochelle
  - Laval
  - Limoges
  - Marseille
  - Montluçon
  - Nice
  - Nîmes
  - Paris
  - Perpignan
  - Poitiers
  - Pringy
  - Rennes
  - Rouen
  - Saint Aubin Sur Cie
  - Saint Julien En Gengvois
  - Saint-Brieuc
  - St-Malo
  - Toulouse
  - Vienne
  - Villeurbanne

REFERENCES:
- [Result] Baulac M, Coulbaut S, Doty P, McShea C, De Backer M, Bartolomei F, Vlaicu M. Adjunctive lacosamide for focal epilepsy: an open-label trial evaluating the impact of flexible titration and dosing on safety and seizure outcomes. Epileptic Disord. 2017 Jun 1;19(2):186-194. doi: 10.1684/epd.2017.0907. PMID 28597842
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a 24-week study, which enrolled 100 patients at 44 sites in France.
Pre-assignment Details: The study comprises a 12-week Titration Phase and a 12-week Maintenance Phase; both phases together are regarded as the 24-week Treatment Period.
  Participant Flow and Baseline Characteristics refer to the Safety Set (SS). The SS includes all subjects that received at least one dose of study medication.
Groups:
- Lacosamide: Flexible dosing between 200 mg/day and 400 mg/day
  Lacosamide : 50 mg tablets bid. Titration phase: (12 weeks) 100 mg/day: duration 1 to 3 weeks. Then uptitration to optimal therapeutic dose of 200 mg/day to 400 mg/day, in steps of 100 mg/day and a time period per step of 1 to 3 weeks.
  Maintenance phase (12 weeks): Optimal therapeutic dose 200 mg/day to 400 mg/day.
  Taper phase if needed: 3 to 4 weeks
Period: Overall Study
Arm/Group | Lacosamide
Started | 100
Completed | 74
Not Completed | 26
Not completed — Adverse Event | 14
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4
Not completed — Lack of Efficacy | 2
Not completed — Other reasons for premature termination | 4

BASELINE CHARACTERISTICS:
Groups:
- Lacosamide: Flexible dosing between 200mg/day and 400mg/day
  Lacosamide: 50 mg tablets bid. Titration phase: (12 weeks) 100 mg/day: duration 1 to 3 weeks. Then uptitration to optimal therapeutic dose of 200 mg/day to 400 mg/day, in steps of 100 mg/day and a time period per step of 1 to 3 weeks.
  Maintenance phase (12 weeks): Optimal therapeutic dose 200 mg/day to 400 mg/day.
  Taper phase if needed: 3 to 4 weeks
Arm/Group | Lacosamide
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 88
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (16.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 45
Region of Enrollment [Number; unit: participants]
  France | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least 1 Treatment-Emergent Adverse Event (TEAE) During the Study
Description: Number of subjects reporting at least 1 Treatment-Emergent Adverse Event (TEAE) during the study. The study is comprised of a 12-week Titration Phase, a 12 -week Maintenance Phase, and a 3 to 4 week Taper Phase if needed.
Time Frame: During the study ( up to 24 - 28 weeks)
Population: Safety Set
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 100
subjects | 64

2. Primary Outcome: Number of Subjects Prematurely Discontinuing Due to a TEAE During the Study
Description: Number of subjects prematurely discontinuing due to a TEAE during the study. The study is comprised of a 12-week Titration Phase, a 12 -week Maintenance Phase, and a 3 to 4 week Taper Phase if needed.
Time Frame: During the study (up to 24 - 28 weeks)
Population: Safety Set
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 100
subjects | 14

3. Secondary Outcome: Percentage of Subjects Retained on Vimpat Through the End of the 24-week Treatment Period
Description: The number of subjects continuing on Vimpat up to and including Visit 4 (Week 24) divided by the number of patients who took at least 1 dose of Vimpat multiplied by 100.
  The overall Treatment Period comprises of a 12-week Titration Phase and 12-week Maintenance Phase.
Time Frame: End of Treatment Period (24-week)
Population: Safety Set
Measure: Number; unit: percentage of subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 100
percentage of subjects | 73

ADVERSE EVENTS:
Time Frame: During the study (up to 24 - 28 weeks). The study is comprised of a 12-week Titration Phase, a 12 -week Maintenance Phase, and a 3 to 4 week Taper Phase if needed.
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 3/100
Other Adverse Events (participants affected / at risk) | 49/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=100)
Diplopia (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=100)
Dizziness (Nervous system disorders) | 42 (46)
Headache (Nervous system disorders) | 8 (9)
Asthenia (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days